CLINICAL TRIAL: NCT07045610
Title: Explore the Primary Resistance Mechanisms of Anaplastic Lymphoma Kinase Inhibitors
Brief Title: Primary Resistance Mechanisms of ALK TKIs
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Director, Head of Surgeon, Principal Investigator, Professor, National Taiwan University Hospital
Other Study IDs: 202504068RINB; TSTS (Other Grant/Funding Number: Taiwan Society of Thoracic Surgeons (TSTS))
Record Dates: First submitted 2025-06-12; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: ALK-positive Advanced NSCLC Patients; Primary Resistance; NGS
Keywords: lung cancer; Anaplastic lymphoma kinase (ALK) gene rearrangement; gene mutation; Primary resistance; Next-generation sequencing; Target therapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The residual lung cancer specimens will be reserved for future lung cancer research and authorize the National Taiwan University Hospital Research Ethics Committee to review whether your consent needs to be re-obtained. The biological specimens will be encoded with a unique number and stored under the control of the National Taiwan University Hospital Ethics Committee in Laboratory 716 on the 7th floor of the National Taiwan University Hospital Research Building for a maximum of 20 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who develop primary resistance or rapid progression after using ALK TKI.: Lung cancer patients who initially use ALK TKI as first-line treatment will be invited to enroll and sign the consent form. Only those who meet the criteria for primary resistance or rapid progression will proceed with tumor sample collection for genetic analysis. Alternatively, patients who develop primary resistance or rapid progression after using ALK TKI and are about to undergo tumor re-biopsy can also sign the subject consent form to be included in this study.
  Interventions: Diagnostic Test: re-biopsy tumor with primary ALK tKI resistance for NGS

INTERVENTIONS:
Diagnostic Test: re-biopsy tumor with primary ALK tKI resistance for NGS — Lung cancer patients who initially use ALK TKI as first-line treatment will be invited to enroll and sign the consent form. Only those who meet the criteria for primary resistance or rapid progression will proceed with tumor sample collection for genetic analysis. Alternatively, patients who develop primary resistance or rapid progression after using ALK TKI and are about to undergo tumor re-biopsy can also sign the subject consent form to be included in this study.

SUMMARY:
Anaplastic lymphoma kinase (ALK) gene rearrangement is a known oncogenic driver in non-small cell lung cancer (NSCLC). ALK tyrosine kinase inhibitors (TKIs) have been clearly shown to produce excellent therapeutic effects and prolong survival in patients with this gene mutation. According to current treatment guidelines, ALK inhibitors are the first-line treatment of choice for ALK-positive advanced NSCLC patients. However, although ALK TKIs are very effective, there is still a small group of patients who do not achieve good treatment outcomes, developing resistance and tumor progression within 3 to 6 months of initial ALK TKI use. This is called primary resistance. Intrinsic resistance to ALK inhibition occurs when the best clinical response after first-generation and second/third-generation TKI treatment is disease progression. Approximately 5-7% of cases after crizotinib treatment, 9% after ceritinib treatment, and 25% after lorlatinib treatment show no response to treatment, and no specific ALK mutation has been found to explain the occurrence of primary resistance. Currently, many different resistance mechanisms are known, some of which are still ALK-related, while others are ALK-independent alternative survival pathways. However, most research focuses on acquired resistance, with very few studies on primary resistance, only a few case reports. Therefore, this study aims to explore the primary ALK TKI resistance mechanisms.

The investigators plan to explore the incidence and mechanisms of primary ALK TKI resistance in ALK-positive advanced NSCLC patients who develop primary resistance or rapid progression (within 3-6 months) during ALK inhibitor treatment by re-obtaining tumor samples for genetic analysis.

DETAILED DESCRIPTION:
Lung cancer is the most common cause of cancer death in Taiwan and worldwide [1]. The traditional chemotherapy, platinum-doublet chemotherapy, provided limited survival benefit. In the recent decades, the major evolution in lung cancer is the molecular subtyping of NSCLC, especially lung adenocarcinoma, which has resulted in a paradigm shift in the management of patients in advanced disease. The target therapy provided better treatment response and longer overall survival. For example, patients with NSCLC harboring Epidermal growth factor receptor (EGFR) mutations can get remarkable benefit and longer survival from EGFR tyrosine kinase inhibitors (TKIs) treatment comparing with the traditional platinum-base chemotherapy [2].

Anaplastic lymphoma kinase (ALK) gene rearrangements define a distinct molecular subset of NSCLC, typically occurring in younger, non-smoking individuals with adenocarcinoma histology [3]. The discovery of ALK fusions, particularly EML4-ALK, revolutionized the treatment of these patients with the development of ALK TKIs. First-generation ALK inhibitors, such as crizotinib, demonstrated remarkable initial responses, significantly improving progression-free survival (PFS) compared to standard chemotherapy [4]. However, the emergence of resistance, both primary and acquired, remains a major clinical challenge.

Primary resistance, defined as the lack of initial response or early progression within the first few months of ALK TKI therapy, occurs in a subset of patients and represents a significant obstacle to optimal treatment outcomes [5]. Primary resistance to ALK inhibition occurs, even with advanced TKI therapies, when the best clinical outcome is disease progression. Notably, approximately 5-7% of patients following crizotinib, 9% following ceritinib, and 25% following lorlatinib demonstrated a lack of response, and in these cases, no identifiable ALK mutations were detected [6]. Unlike acquired resistance, which typically arises from secondary mutations within the ALK kinase domain or activation of bypass signaling pathways, the mechanisms underlying primary resistance are less well understood.

Several potential factors contribute to primary resistance. One key aspect involves inherent tumor heterogeneity. NSCLC tumors are complex ecosystems with diverse subclones, some of which may harbor pre-existing genetic alterations that confer resistance to ALK inhibition [7]. These alterations might include co-occurring mutations in genes involved in cell signaling pathways, such as KRAS, EGFR, or TP53, which can bypass ALK dependence [6]. Furthermore, variations in ALK fusion isoforms or copy number alterations may also influence initial drug sensitivity. For example, some less common ALK fusion variants might possess distinct structural properties that reduce their affinity for ALK TKIs.

Another potential mechanism involves the tumor microenvironment (TME). The TME, composed of stromal cells, immune cells, and extracellular matrix, plays a critical role in tumor growth and drug response [8]. Components of the TME, such as cancer-associated fibroblasts (CAFs) and immunosuppressive cells, can secrete growth factors and cytokines that activate alternative signaling pathways, thereby promoting resistance to ALK inhibition. Additionally, the TME can create a physical barrier that limits drug penetration and efficacy.

Furthermore, the complexity of ALK signaling networks and the potential for activation of bypass pathways contribute to primary resistance. For example, activation of the EGFR or MET signaling pathways can provide alternative growth signals, bypassing the need for ALK activation [9]. Understanding these bypass pathways is crucial for developing combination therapies that can overcome primary resistance.

Investigating primary resistance requires a comprehensive approach that integrates genomic, transcriptomic, and proteomic analyses. Next-generation sequencing (NGS) can identify pre-existing genetic alterations that confer resistance. Single-cell RNA sequencing can dissect tumor heterogeneity and identify resistant subclones. Proteomic profiling can reveal activation of bypass signaling pathways. Clinical studies analyzing pre-treatment tumor samples and correlating genomic and clinical data are essential for identifying predictive biomarkers of primary resistance.

In summary, primary resistance to ALK TKIs in NSCLC is a complex phenomenon driven by multiple factors, including tumor heterogeneity, TME interactions, pharmacokinetic variations, and activation of bypass signaling pathways. Further research is needed to elucidate the precise mechanisms underlying primary resistance and to develop strategies to overcome this clinical challenge, ultimately improving outcomes for patients with ALK-positive NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Histologically or cytologically diagnosed NSCLC
3. ALK gene fusion detected at initial diagnosis of NSCLC
4. Patients exhibiting primary resistance to ALK-TKI therapy, defined as the absence of initial response or progression within 3 to 6 months of treatment initiation, were included.
5. Able and willing to provide written informed consent prior to performing any study related procedures and to comply with the study protocol.

Exclusion Criteria:

1. Unable to provide written inform consent
2. The patients had received other systemic treatments except ALK TKI.
3. Unable to undergo tumor biopsy or venipuncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALK-positive advanced NSCLC patients who develop primary resistance or rapid progression (within 3-6 months) during ALK inhibitor treatment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
resistance mechanism | From ALK TKI treatment to primary resistance or rapid progression for less than 6 months.
  Lung cancer patients who initially use ALK TKI as first-line treatment will be invited to enroll and sign the consent form. Only those who meet the criteria for primary resistance or rapid progression will proceed with tumor sample collection for NGS analysis. Alternatively, patients who develop primary resistance or rapid progression after using ALK TKI and are about to undergo tumor re-biopsy can also sign the subject consent form to be included in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Shing Chen, Professor, Principal Investigator — Taiwan Society of Thoracic Surgeons
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoda S, Lin JJ, Lawrence MS, Burke BJ, Friboulet L, Langenbucher A, Dardaei L, Prutisto-Chang K, Dagogo-Jack I, Timofeevski S, Hubbeling H, Gainor JF, Ferris LA, Riley AK, Kattermann KE, Timonina D, Heist RS, Iafrate AJ, Benes CH, Lennerz JK, Mino-Kenudson M, Engelman JA, Johnson TW, Hata AN, Shaw AT. Sequential ALK Inhibitors Can Select for Lorlatinib-Resistant Compound ALK Mutations in ALK-Positive Lung Cancer. Cancer Discov. 2018 Jun;8(6):714-729. doi: 10.1158/2159-8290.CD-17-1256. Epub 2018 Apr 12. PMID 29650534
- [Background] Shaw AT, Kim DW, Mehra R, Tan DS, Felip E, Chow LQ, Camidge DR, Vansteenkiste J, Sharma S, De Pas T, Riely GJ, Solomon BJ, Wolf J, Thomas M, Schuler M, Liu G, Santoro A, Lau YY, Goldwasser M, Boral AL, Engelman JA. Ceritinib in ALK-rearranged non-small-cell lung cancer. N Engl J Med. 2014 Mar 27;370(13):1189-97. doi: 10.1056/NEJMoa1311107. PMID 24670165
- [Background] Hinshaw DC, Shevde LA. The Tumor Microenvironment Innately Modulates Cancer Progression. Cancer Res. 2019 Sep 15;79(18):4557-4566. doi: 10.1158/0008-5472.CAN-18-3962. Epub 2019 Jul 26. PMID 31350295
- [Background] Jamal-Hanjani M, Wilson GA, McGranahan N, Birkbak NJ, Watkins TBK, Veeriah S, Shafi S, Johnson DH, Mitter R, Rosenthal R, Salm M, Horswell S, Escudero M, Matthews N, Rowan A, Chambers T, Moore DA, Turajlic S, Xu H, Lee SM, Forster MD, Ahmad T, Hiley CT, Abbosh C, Falzon M, Borg E, Marafioti T, Lawrence D, Hayward M, Kolvekar S, Panagiotopoulos N, Janes SM, Thakrar R, Ahmed A, Blackhall F, Summers Y, Shah R, Joseph L, Quinn AM, Crosbie PA, Naidu B, Middleton G, Langman G, Trotter S, Nicolson M, Remmen H, Kerr K, Chetty M, Gomersall L, Fennell DA, Nakas A, Rathinam S, Anand G, Khan S, Russell P, Ezhil V, Ismail B, Irvin-Sellers M, Prakash V, Lester JF, Kornaszewska M, Attanoos R, Adams H, Davies H, Dentro S, Taniere P, O'Sullivan B, Lowe HL, Hartley JA, Iles N, Bell H, Ngai Y, Shaw JA, Herrero J, Szallasi Z, Schwarz RF, Stewart A, Quezada SA, Le Quesne J, Van Loo P, Dive C, Hackshaw A, Swanton C; TRACERx Consortium. Tracking the Evolution of Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Jun 1;376(22):2109-2121. doi: 10.1056/NEJMoa1616288. Epub 2017 Apr 26. PMID 28445112
- [Background] Gainor JF, Dardaei L, Yoda S, Friboulet L, Leshchiner I, Katayama R, Dagogo-Jack I, Gadgeel S, Schultz K, Singh M, Chin E, Parks M, Lee D, DiCecca RH, Lockerman E, Huynh T, Logan J, Ritterhouse LL, Le LP, Muniappan A, Digumarthy S, Channick C, Keyes C, Getz G, Dias-Santagata D, Heist RS, Lennerz J, Sequist LV, Benes CH, Iafrate AJ, Mino-Kenudson M, Engelman JA, Shaw AT. Molecular Mechanisms of Resistance to First- and Second-Generation ALK Inhibitors in ALK-Rearranged Lung Cancer. Cancer Discov. 2016 Oct;6(10):1118-1133. doi: 10.1158/2159-8290.CD-16-0596. Epub 2016 Jul 18. PMID 27432227
- [Background] Katayama R, Shaw AT, Khan TM, Mino-Kenudson M, Solomon BJ, Halmos B, Jessop NA, Wain JC, Yeo AT, Benes C, Drew L, Saeh JC, Crosby K, Sequist LV, Iafrate AJ, Engelman JA. Mechanisms of acquired crizotinib resistance in ALK-rearranged lung Cancers. Sci Transl Med. 2012 Feb 8;4(120):120ra17. doi: 10.1126/scitranslmed.3003316. Epub 2012 Jan 25. PMID 22277784
- [Background] Camidge DR, Bang YJ, Kwak EL, Iafrate AJ, Varella-Garcia M, Fox SB, Riely GJ, Solomon B, Ou SH, Kim DW, Salgia R, Fidias P, Engelman JA, Gandhi L, Janne PA, Costa DB, Shapiro GI, Lorusso P, Ruffner K, Stephenson P, Tang Y, Wilner K, Clark JW, Shaw AT. Activity and safety of crizotinib in patients with ALK-positive non-small-cell lung cancer: updated results from a phase 1 study. Lancet Oncol. 2012 Oct;13(10):1011-9. doi: 10.1016/S1470-2045(12)70344-3. Epub 2012 Sep 4. PMID 22954507
- [Background] Shaw AT, Yeap BY, Mino-Kenudson M, Digumarthy SR, Costa DB, Heist RS, Solomon B, Stubbs H, Admane S, McDermott U, Settleman J, Kobayashi S, Mark EJ, Rodig SJ, Chirieac LR, Kwak EL, Lynch TJ, Iafrate AJ. Clinical features and outcome of patients with non-small-cell lung cancer who harbor EML4-ALK. J Clin Oncol. 2009 Sep 10;27(26):4247-53. doi: 10.1200/JCO.2009.22.6993. Epub 2009 Aug 10. PMID 19667264
- [Background] Lynch TJ, Bell DW, Sordella R, Gurubhagavatula S, Okimoto RA, Brannigan BW, Harris PL, Haserlat SM, Supko JG, Haluska FG, Louis DN, Christiani DC, Settleman J, Haber DA. Activating mutations in the epidermal growth factor receptor underlying responsiveness of non-small-cell lung cancer to gefitinib. N Engl J Med. 2004 May 20;350(21):2129-39. doi: 10.1056/NEJMoa040938. Epub 2004 Apr 29. PMID 15118073
- [Background] Siegel RL, Kratzer TB, Giaquinto AN, Sung H, Jemal A. Cancer statistics, 2025. CA Cancer J Clin. 2025 Jan-Feb;75(1):10-45. doi: 10.3322/caac.21871. Epub 2025 Jan 16. PMID 39817679

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT07045610/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT07045610/ICF_001.pdf